CLINICAL TRIAL: NCT05140174
Title: Incorporating Radical Healing and Addressing Internalized Transnegativity in Psychotherapy for Transgender, Two-Spirit, and Nonbinary People of Color: An Open Clinical Trial
Brief Title: Psychotherapy Interventions to Support Transgender, Two-Spirit, and Nonbinary People of Color
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-1133; A171600 (Other: UW Madison); Protocol Version 12/1/2021 (Other: UW Madison)
Record Dates: First submitted 2021-11-17; First posted 2021-12-01 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Mental Health
Keywords: mental health care; training; transgender; nonbinary; two spirit; access
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: Uncontrolled psychotherapy trial (longitudinal study with no control group)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- RHIS Informed Psychotherapy (Experimental): Therapists will be trained in Radical Healing and Internalized Stigma (RHIS) and meet with their clients as part of their usual care for 15 tele-psychotherapy sessions
  Interventions: Other: Radical Healing and Internalized Stigma (RHIS) Training

INTERVENTIONS:
Other: Radical Healing and Internalized Stigma (RHIS) Training — 8-hour RHIS training includes, readings that discuss radical healing and internalized stigma, access to didactic information regarding radical healing and internalized stigma. Therapists will role play certain scenarios that may involve minority stress experiences and discuss with the trainers different types of responses that could be therapeutic. The training will focus on the most up to date research regarding transgender mental health, minority stress, radical healing, and role-plays that focus on these processes.

SUMMARY:
The proposed research will use a community-based participatory research (CBPR) approach to engage with community organizations to design and implement a project that trains therapists to provide effective, supportive, and engaged therapy to two-spirit, transgender, and nonbinary (2STNB) clients most impacted by barriers in accessing mental health care. 10 2STNB licensed mental health therapists will be identified and 50 2STNB of their clients will be enrolled and can expect to be on study for 10-20 months.

DETAILED DESCRIPTION:
The long-term aim of this research is to ensure that therapists have access to training and engage in effective psychotherapy that ultimately reaches Two-spirit, transgender, and nonbinary (2STNB) clients who are the most impacted by unequal systems that create mental health concerns. To make real improvement in reaching TNB populations who lack the most access to mental health care, therapists must be properly trained and data from clients about their mental health experiences must be obtained. The proposed research will use a community-based participatory research (CBPR) approach to engage with community organizations to design and implement a project that trains therapists to provide effective, supportive, and engaged therapy to TNB clients most impacted by barriers in accessing mental health care.

Intervention:

* Therapist Training: The Radical Healing and Internalized Stigma (RHIS) training provides education to therapists on radical healing and internalized stress. The ten therapists employed by the study will engage in an 8 hour intensive training by consultants hired to be on this study.
* Participants:

  * T0 - baseline surveys
  * T1a to T1p - psychotherapy sessions (session complete within 11 months)
  * T2 - end intervention surveys
  * T3 - post intervention follow up (up to 6 months post intervention)

Aim 1: Determine best methods for recruiting 2STNB clients (e.g., increasing access to care), with attention to specific populations and barriers (BIPOC, lack of trust, finances, identity match, etc.)

Aim 2: Examine the feasibility/acceptability of a specialized training for therapists that focuses on healing and internalized stigma

Aim 3: Longitudinally investigate the impact of access to mental health care (e-therapy) on 2STNB people's well-being/mental health.

Endpoints:

The primary endpoint of the study is to determine if the study actually improved access to mental health care for study participants--this will be determined through qualitative interviewing. An additional endpoint is determining feasibility/acceptability of the study, which will also be assessed via qualitative methods.

A secondary endpoint for this study will be to determine if clients experienced psychological improvement in their mental health over the course of the study.

ELIGIBILITY:
Inclusion Criteria:

* fluent in written and spoken English and/or Spanish
* willingness to participate in pre/ post/ session-by session assessments and 15 individual psychotherapy treatment sessions
* individual identifies as transgender, Two-Spirit, or nonbinary (or somewhere along the gender minority spectrum)
* individual identifies as Black, Indigenous/Native, or otherwise as a person of color
* not currently in individual therapy with another therapist

Exclusion Criteria:

* reports current, unmanaged serious/persistent mental health symptoms requiring inpatient treatment (e.g., hallucinations, delusions)
* individual does not identify as transgender, Two-Spirit, or nonbinary (or somewhere along the gender minority spectrum)
* currently in therapy with an individual therapist

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Participants identify as transgender, Two-Spirit, or nonbinary (or somewhere along the gender minority spectrum) and identifies as Black, Indigenous/Native, or otherwise as a person of color.
Enrollment: 51 (Actual)
Dates: Start 2022-01-14 (Actual); Primary Completion 2023-08-10 (Actual); Study Completion 2023-08-10 (Actual)

PRIMARY OUTCOMES:
Number of Participants who Find the Intervention Acceptable | up to 20 months
  Acceptability of the Intervention will be assessed qualitatively via semi-structured interviews post intervention.
Number of Participants Who Find Intervention Feasible | up to 20 months
  Feasibility of the Intervention will be assessed qualitatively via semi-structured interviews post intervention.
Number of Participants Who Indicate Barriers to Therapy Were Decreased | up to 20 months
  Participant Satisfaction with RHIS Intervention will be assessed qualitatively by semi-structured interview with researcher where access to mental health will be queried.

SECONDARY OUTCOMES:
Change in Percent "Yes" on Yes/No subscales on Gender Minority Stress and Resilience Measure (GMSR) | baseline, post-intervention (up to 14 months), follow-up (up to 20 months)
  Designed for use with transgender, nonbinary, and gender nonconforming people, the GMSR measure is one of the few that assesses gender identity-related constructs. It was designed to take into account unique gender minority stressors, such as internalized transphobia, and concealment of identity, and resilience factors including community connectedness and pride. The first 3 sub-scales for gender-related discrimination, gender-related rejection, and gender-related victimization are yes/no responses, where 'yes' responses indicated gender-related discrimination, rejection, and victimization.
Change in Gender Minority Stress and Resilience Measure (GMSR) Scores | baseline, post-intervention (up to 14 months), follow-up (up to 20 months)
  Designed for use with transgender, nonbinary, and gender nonconforming people, the GMSR measure is one of the few that assesses gender identity-related constructs. It was designed to take into account unique gender minority stressors, such as internalized transphobia, and concealment of identity, and resilience factors including community connectedness and pride. The last sub-scales are given on a 5-point Likert response scale (Strongly Disagree = 0 to Strongly Agree = 4) and responses are summed. Higher scores are indicative of greater phenomena. Sub-scales are as follows:
  * Non-Affirmation: 6-items (0-24)
  * Internalized Transphobia: 8-items (0-32)
  * Pride: 8-items (0-32)
  * Negative Expectations for Future Events: 9-items (0-36)
  * Non-Disclosure: 5-items (0-20)
  * Community Connectedness: 5-items (0-20)
Change in Outcome Questionnaire-45 (OQ-45) Score | baseline, post-intervention (up to 14 months), follow-up (up to 20 months)
  The OQ-45 is a measure of how a person has felt in the past week. Total possible range of scores from 0-180, where the higher the score, the more disturbed the participant.
Change in Depression, Anxiety, and Stress Scale (DASS) Scores | baseline, post-intervention (up to 14 months), follow-up (up to 20 months)
  The DASS is a measure of how perceived depression, anxiety, and stress in the past week. Total possible range of scores for each domain is 0-21, where higher scores indicate more severe depression, anxiety, and stress.
Change in Coping with Discrimination Scale (CDS) Score | baseline, post-intervention (up to 14 months), follow-up (up to 20 months)
  CDS is a 25-item scale measuring five specific strategies (i.e., education/advocacy, internalization, drug and alcohol use, resistance, and detachment) that minority individuals may use when coping with experiences of prejudice and discrimination. Items are responded to on a 6-point Likert-type scale ranging from 1 = never like me to 6 = always like me, for a range of 25 - 150. The investigators will analyze a longitudinal change through time, where better coping is evidenced by higher scores.
Change in Schwartz Outcome Scale Score | baseline, post-intervention (up to 14 months), follow-up (up to 20 months)
  This is a 10-item measure of how someone feels over the previous 7 days. Total possible range of scores is 0-100 where higher scores indicate improved outcome.
Change in Client Task Specific Change Measure | baseline, post-intervention (up to 14 months), follow-up (up to 20 months)
  This is a 16-item measure of how someone feels they've changed. Total possible range of scores is 16-112, where higher scores indicate improved outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Budge, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Budge SL, Ben L, Lynn S, Tebbe EA. A Thematic Analysis of Teletherapy Benefits and Challenges for Two Spirit, Transgender, and Nonbinary People of Color: Qualitative Results from the HOPE Trial. Telemed J E Health. 2025 Nov 21. doi: 10.1177/15305627251399268. Online ahead of print. PMID 41313600